CLINICAL TRIAL: NCT05236829
Title: Comparison of Exercise Capacity, Physical Activity Level and Quality of Life in Prolactinoma Patients and Healthy Individuals
Brief Title: Exercise Capacity and Physical Activity Level in Prolactinoma Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO21/728
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prolactinoma
Keywords: Prolactinoma; exercise capacity; physical activity; quality of life
MeSH Terms: conditions — Prolactinoma; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Healthy women aged 18-55 who have not been diagnosed with any chronic disease and pituitary adenoma
- Patient with Prolactinoma group: Women between the ages of 18-55 diagnosed with Prolactinoma

SUMMARY:
Prolactinoma, one of the most common pituitary adenomas, is an adenoma that causes excessive prolactin (PRL) secretion. An increase in prolactin level can cause weakness, decrease in muscle mass and fatigue. It is not known in detail to what extent it affects quality of life, functional exercise capacity, cardiovascular disease risk factors, physical activity level, fatigue and sleep quality in prolactinoma patients. It is aimed to compare how much exercise capacity, physical activity level, sleep quality, perception of fatigue and quality of life of prolactinoma patients are affected compared to healthy individuals and to examine the factors associated with exercise capacity in prolactinoma patients.

DETAILED DESCRIPTION:
Prolactinoma is a pituitary adenoma caused by excessive prolactin secretion. More than 70% of patients are women. Many physiological conditions such as pregnancy, breastfeeding, breast stimulation, stress, exercise and sleep can also increase PRL levels. Prolactin can affect arterial stiffness and blood pressure and cause atherosclerosis in early menopause. In addition to these, it has negative effects on heart rhythm and heart failure. In addition to these clinical findings, the extent to which body weight gain and fatigue symptoms affect quality of life, functional exercise capacity, cardiovascular disease risk factors, physical activity level, fatigue and sleep quality in prolactinoma patients is not known in detail. There are very few studies on these subjects. Height, weight, waist circumference, hip circumference will be measured for all participants, waist-hip ratio and body mass index (BMI) will be calculated. The exercise capacity levels of the individuals who will participate in the study will be evaluated with the 6 Minute Walk Test (6MWT). Risk factors knowledge levels about cardiovascular diseases will be evaluated with Cardiovascular Diseases Risk Factors Knowledge Level (CARRIF-BD) Scale. Physical activity level will be evaluated with the Turkish version of the short form of the International Physical Activity Questionnaire (IPAQ). The Pittsburgh Sleep Quality Index (PUKI) was used to evaluate sleep quality. Fatigue assessment will be evaluated with the Multidimensional Fatigue Rating Scale. quality of life will be evaluated with the SF-36 short form. Measurement of knee extensor muscle strength will be made with a portable digital dynamometer (JTECH, Medical Commander Powertrack II, Midvale, USA). Peripheral muscle endurance assessment will be done by bilateral squat test.

ELIGIBILITY:
Inclusion Criteria of patients:

* Being between the ages of 18-55
* Woman
* Being diagnosed with prolactinoma
* Volunteering to participate in the study

Exclusion Criteria of the patients :

* Patients with neurological, cognitive or orthopedic disease that will affect the measurements
* Patients with severe respiratory disease (FEV1 < 35%; FVC < 50%)
* Presence of acute infection
* Presence of malignancy
* Presence of dementia
* Patients who have had a cardiovascular event in the last 6 months
* Less than 50% of the ejection fraction
* Patients with uncontrolled hypertension
* Individuals with a diagnosis of uncontrolled diabetes mellitus will not be included in the study.

Healthy group inclusion criteria:

* Being between the ages of 18-55
* Woman
* Not being diagnosed with any pituitary adenoma
* Volunteering to participate in the study

Healthy group exclusion criteria:

* Cases with neurological, cognitive or orthopedic diseases that will affect the measurements
* Cases with severe respiratory disease (FEV1 < 35%; FVC < 50%)
* Presence of acute infection
* Presence of malignancy
* Presence of dementia
* Cases who have had a cardiovascular event in the last 6 months
* Less than 50% of the ejection fraction
* Patients with uncontrolled hypertension
* Cases with uncontrolled diabetes mellitus diagnosis will not be included in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy group: Individuals between the ages of 18-55, female, not diagnosed with a pituitary adenoma, volunteered to participate in the study.
  Patient group: Individuals aged 18-55, female, diagnosed with prolactinoma, volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Aerobic Exercise Capacity | day 1
  Exercise capacity levels of individuals will be evaluated with the 6-Minute Walking Test (6MWT).
Physical Activity Level | day 1
  Physical activity level will be evaluated with the Turkish version of the short form of the International Physical Activity Questionnaire (IPAQ). The scale consists of 7 questions. Activities and sitting time in the last 1 week are recorded in minutes.
Life quality | day 1
  The Pittsburgh Sleep Quality Index (PUKI) will be used to assess sleep quality. The scale has eight sub-parameters and consists of 36 items. Scoring is between 0 and 100. Higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Peripheral Muscle Strength | day 1
  Knee extensor muscle strength will be measured in individuals in sitting position and knee extension. 3 repetitions will be applied for the right and left sides and the results will be recorded in kilograms.
Peripheral Muscle Endurance | day 1
  Evaluation will be done with bilateral squat test. Participants initially stand with hips and shoulders in line, knees fully extended, then squat with knees flexed to 90°, then return to starting position. The exact number of repetitions performed in 30 seconds is recorded.
Cardiovascular Diseases Risk Factors Knowledge Level | day 1
  Individuals' knowledge of risk factors about cardiovascular diseases will be evaluated with the Cardiovascular Diseases Risk Factors Knowledge Level (CARRIF-BD) Scale. The scale consists of 28 items. It is concluded that the higher the scale score, the higher the level of knowledge of the individual.
Fatigue perception | day 1
  Individuals' fatigue perception will be assessed by Multidimensional Assessment of Fatigue (MAF) Scale. The scores to be taken from the scale vary between 1-50. As the scores increase, the level of fatigue also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Erkoc A, Eroglu I, Erbas T, Kutukcu EC. Muscle function, exercise capacity, physical activity level and cardiovascular disease risk factor knowledge in patients with prolactinoma. Endocrine. 2024 Sep;85(3):1337-1345. doi: 10.1007/s12020-024-03880-7. Epub 2024 May 27. PMID 38801597